CLINICAL TRIAL: NCT04632706
Title: A Randomised, Double-Blind, Placebo-Controlled, Exploratory Phase I Trial Assessing the Pharmacokinetic Profile, Safety and Tolerability of a Continuous Daily Dosing Regimen of Active IMP in Healthy Volunteers
Brief Title: Exploratory Ph I Trial of the Active IMP in Healthy Volunteers in Relation to COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedinCell S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: mdc-TTG-CT-001
Record Dates: First submitted 2020-10-26; First posted 2020-11-17 (Actual); Results first posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: The study is a placebo-controlled, double-blinded exploratory study to investigate safety, Pk and tolerability of a continuous daily dosing of the active drugs (at 3 different doses) in healthy participants.
Who Masked: Participant, Investigator
Masking Description: The study is double-blinded. Patients will be randomised to receive 1 of 3 doses of the Active IMP or a matching placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 50mcg/kg (oral) (Experimental): Ivermectin loading dose of 200 mcg/kg followed by daily doses of 50mcg/kg from D2 to D28
  Interventions: Drug: Ivermectin
- 75mcg/kg (oral) (Experimental): Ivermectin loading dose of 200 mcg/kg followed by daily doses of 75mcg/kg from D2 to D28
  Interventions: Drug: Ivermectin
- 100mcg/kg (oral) (Experimental): Ivermectin loading dose of 200 mcg/kg followed by daily doses of 100mcg/kg from D2 to D28
  Interventions: Drug: Ivermectin
- Matching Placebo (oral) (Placebo Comparator): Placebo using tablets identical to the Active IMP
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — Ivermectin: Investigation of the safety, tolerability and the pharmacokinetic profile of the active IMP in an exploratory study
  Arms: 100mcg/kg (oral); 50mcg/kg (oral); 75mcg/kg (oral)
Drug: Placebo — Matching Placebo to the Active IMP.
  Arms: Matching Placebo (oral)

SUMMARY:
An early stage trial to check how safe and tolerable, as well as how the body handles continuous daily use of Active IMP over 28 days in healthy volunteers.

DETAILED DESCRIPTION:
Detailed information restricted because this is a Phase 1 clinical trial.

ELIGIBILITY:
Important Inclusion Criteria:

* Subject is male of any ethnic origin.
* Subject is aged between 18 to 45 years, inclusive.
* Subject has a body mass index (BMI) of 18.5 to 32.0 kg/m2, inclusive.
* Subject is ≥50 kg.
* Negative reverse transcription polymerase chain reaction (RT-PCR) Test for severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) at Screening and negative lateral flow immunoassay test for SARS-CoV-2 at Day -1.
* Healthy as determined by a responsible physician, based on medical evaluation including medical history, physical examinations, neurological examinations, concomitant medication, vital signs, 12-lead ECG and clinical laboratory evaluations.
* Male subjects must use a condom during the study and for 3 months after their final dose of study medication, if their partner is a woman of childbearing potential. In addition, their female partner of childbearing potential must use an additional method of highly effective contraception from first dosing until 3 months following final dosing.

Important Exclusion Criteria:

* Clinically relevant history of abnormal physical or mental health (defined as any subject requiring medical, psychological or pharmacotherapeutic intervention for mental illness) interfering with the study as determined by medical history and physical examinations obtained during Screening and Day -1 as judged by the Investigator (including [but not limited to], neurological, psychiatric, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder).
* Any other concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study as outlined in this Protocol, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
* Evidence of previous SARS-CoV-2 infection from medical history.
* Ophthalmologic disorder (moderate and sever retina or optic nerve pathology; cataracts excluded).
* Subjects with a diagnosis of asthma or any other respiratory conditions.
* A neurologic disorder that may compromise blood brain barrier permeability (stroke within 90 days, brain tumour, multiple sclerosis, or other neuroinflammatory condition, a neurodegenerative disorder, epilepsy) or history of seizures.
* Positive test for hepatitis B surface antigen (HBsAg), anti-hepatitis C antibody (anti-HCV) or human immunodeficiency virus I and II (anti-HIV I/II) at Screening.
* The subject has participated in a clinical study and has received a medication or a new chemical entity within 3 months or 5 half-lives (whichever is longer) prior to first dosing of current study medication.
* Use of any drugs that are known substrates of CYP3A4, P-glycoprotein (P-gp) from within 4 weeks of Screening and unable to refrain from them until the end of the study (e.g., rifampicin, quinidine, amiodarone, diltiazem, spironolactone, verapamil, clarithromycin, erythromycin, itraconazole, ketoconazole, cyclosporine, tacrolimus, indinavir, ritonavir or cobicistat). Use of critical CYP3A4 substrate drugs such as warfarin or coumarin anticoagulants.
* Recent or expected microfilaricidal drug use, including ivermectin, or travel history to areas that are endemic for Loa loa or onchocerciasis (Angola, Cameroon, Central African Republic, Chad, Democratic Republic of Congo, Ethiopia, Equatorial, Guinea, Gabon, Republic of Congo, Nigeria and Sudan).
* Use of medications having potential activity against SARS-CoV-2 such as hydroxychloroquine, chloroquine, lopinavir, ritonavir, remdesivir, azithromycin, in the 30 days prior to Screening and unable to refrain from them until the end of the study.
* Consumption of any food or drinks containing cranberry, pomegranate, starfruit, grapefruit, pomelos, exotic citrus fruits or Seville oranges (including marmalade and juices made from these fruits) within 14 days prior to first dosing until the end of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pui Man Leung, MD, Principal Investigator — MAC Clinical Research
Locations (1):
- MAC Clinical Research Manchester (Early Phase Unit), Neuroscience Centre of Excellence, Manchester, Greater Mancherster, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Matching Placebo (Oral): Placebo tablets matching the Active Investigative Medicinal Product (IMP)
Period: Overall Study
Arm/Group | 50mcg/kg (Oral) | 75mcg/kg (Oral) | 100mcg/kg (Oral) | Matching Placebo (Oral)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Matching Placebo (Oral): Placebo tablets matching the Active IMP
- Total: Total of all reporting groups
Arm/Group | 50mcg/kg (Oral) | 75mcg/kg (Oral) | 100mcg/kg (Oral) | Matching Placebo (Oral) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Full Range); unit: years] | 35.2 [25 to 45] | 29.3 [21 to 43] | 30.3 [21 to 43] | 28.2 [23 to 35] | 30.8 [21 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 6 | 6 | 24
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 24.95 [19.43 to 30.85] | 25.79 [21.73 to 29.24] | 25.84 [20.04 to 31.65] | 25.57 [23.57 to 29.10] | 25.54 [19.43 to 31.65]

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Concentrations - (Maximum Plasma Concentration [Cmax])
Description: Maximum plasma concentration (Cmax)
Time Frame: D1, D2 and D28
Population: All 18 participants on active IMP were eligible and analyzed for this endpoint. Number Analyzed per Row represents those with data available at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 50mcg/kg (Oral) | 75mcg/kg (Oral) | 100mcg/kg (Oral)
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Day 1 after loading dose of 200mcg/kg (oral) for all active treatment groups | 57.2 (28.9) | 41.7 (73.5) | 46.5 (53.6)
  Day 2 (first day on respective dose of active treatment) | 22.3 (32.5) | 24.4 (42.5) | 33.2 (62.6)
  Day 28 (last day of active treatment): number analyzed (Participants) | 6 | 6 | 5
  Day 28 (last day of active treatment) | 23.3 (52.8) | 31.9 (27.6) | 44.4 (68.8)
Statistical Analysis 1: Comparison: 50mcg/kg (Oral) vs 75mcg/kg (Oral) vs 100mcg/kg (Oral); Assessment of dose proportionality on D2 and D28; Test type: Other; p = 0.803, Mixed Models Analysis — If the p-value is more than 0.05 then dose proportionality can not be confirmed

2. Primary Outcome: Pharmacokinetic Concentrations - (Time to Reach Cmax [Tmax])
Description: Time to reach Cmax (Tmax)
Time Frame: D1, D2 and D28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | 50mcg/kg (Oral) | 75mcg/kg (Oral) | 100mcg/kg (Oral)
Number analyzed (Participants) | 6 | 6 | 6
hr
  Day 1 after loading dose of 200mcg/kg (oral) for all active treatment groups | 2.53 (36.8) | 3.03 (50.6) | 4.8 (47.2)
  Day 2 (first day on respective dose of active treatment) | 3.82 (36.7) | 2.85 (38.8) | 3.23 (34.5)
  Day 28 (last day of active treatment): number analyzed (Participants) | 6 | 6 | 5
  Day 28 (last day of active treatment) | 2.83 (39.2) | 3.03 (50.7) | 3.03 (39.4)

3. Primary Outcome: Pharmacokinetic Concentrations - (Area Under the Plasma Concentration-time Curve From Zero to 24 Hours [AUC0-24hr])
Description: area under the plasma concentration-time curve from zero to 24 hours (AUC0-24hr) concentration-time curve from zero to 24 hours (AUC0-24hr)
Time Frame: D1, D2 and D28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 50mcg/kg (Oral) | 75mcg/kg (Oral) | 100mcg/kg (Oral)
Number analyzed (Participants) | 6 | 6 | 6
ng*h/mL
  Day 1 after loading dose of 200mcg/kg (oral) for all active treatment groups | 568 (33.6) | 449 (62.0) | 523 (60.5)
  Day 2 (first day on respective dose of active treatment) | 906 (31.4) | 779 (53.1) | 941 (59.0)
  Day 28 (last day of active treatment): number analyzed (Participants) | 6 | 6 | 5
  Day 28 (last day of active treatment) | 1.06 (36.6) | 1.5 (47.5) | 1.75 (20.6)
Statistical Analysis 1: Comparison: 50mcg/kg (Oral) vs 75mcg/kg (Oral) vs 100mcg/kg (Oral); Assessment of dose proportionality on D2 and D28; Test type: Other; p = 0.689, Mixed Models Analysis — If the p-value is more than 0.05 then dose proportionality can not be confirmed

4. Primary Outcome: Pharmacokinetic Concentrations - (Apparent Terminal Half-Life [T1/2])
Description: apparent terminal half-life (t1/2)
Time Frame: D28
Population: 17 participants on active IMP were analysed for this endpoint. On day 21 one subject in the 100 μg/kg/day ivermectin treatment group was discontinued.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | 50mcg/kg (Oral) | 75mcg/kg (Oral) | 100mcg/kg (Oral)
Number analyzed (Participants) | 6 | 6 | 5
hr | 102 (60.1) | 99.2 (47.3) | 127 (47.2)

5. Secondary Outcome: Safety and Tolerability - Treatment Emergent Adverse Events (TEAEs)
Description: Clinical safety data from adverse event (AE) reporting
Time Frame: From Screening (Day -28) to Follow up visit (Day +42) plus 7 additional days.
Population: All 24 included participants were eligible and analysed for this endpoint
Measure: Number; unit: TEAE
Arm/Group | 50mcg/kg (Oral) | 75mcg/kg (Oral) | 100mcg/kg (Oral) | Matching Placebo (Oral)
Number analyzed (Participants) | 6 | 6 | 6 | 6
TEAE
  Any TEAE | 24 | 5 | 2 | 21
  Any serious TEAE | 0 | 0 | 0 | 0
  Any TEAE leading to discontinuation - due to Study Medication-related TEAE | 0 | 0 | 0 | 0
  Any TEAE leading to discontinuation - other reason | 0 | 0 | 1 | 0
  TEAE - mild severity | 24 | 5 | 2 | 20
  TEAE - moderate severity | 0 | 0 | 0 | 1
  Causality (All TEAEs) - Not related | 21 | 3 | 2 | 20
  Causality (All TEAEs) - Related (possibly and probably) | 3 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: From Screening (Day -28) to Follow up visit (Day +42) plus 7 additional days
Groups:
- Ivermectin Overall: Ivermectin loading dose of 200 mcg/kg followed by daily doses of either 50, 75, or 100mcg/kg from D2 to D28.
- Total (Ivermectin Overall and Placebo): All study participants
Arm/Group | 50mcg/kg (Oral) | 75mcg/kg (Oral) | 100mcg/kg (Oral) | Matching Placebo (Oral) | Ivermectin Overall | Total (Ivermectin Overall and Placebo)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/18 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/18 | 0/24
Other Adverse Events (participants affected / at risk) | 6/6 | 3/6 | 2/6 | 6/6 | 11/18 | 17/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mcg/kg (Oral) (N=6) | 75mcg/kg (Oral) (N=6) | 100mcg/kg (Oral) (N=6) | Matching Placebo (Oral) (N=6) | Ivermectin Overall (N=18) | Total (Ivermectin Overall and Placebo) (N=24)
Palpitations (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (3) — 2 subjects on active treatment experienced 3 AEs; 2 AEs (one in each subject) were possibly related to study drug
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — 1 subject on active treatment experienced 1 AE; it was possibly related to the study drug
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 4 (5) — 3 subjects on active treatment experienced 4 AEs and 1 subject on placebo experienced 1 AE; 1 AE in the treatment group was possibly related to the study drug
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) — 1 subject on placebo experienced 2 AEs
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — 1 subject on active treatment experienced 1 AE; it was not related to the study drug
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — 1 subject on active treatment experienced 1 AE; it was not related to the study drug
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — 1 subject on active treatment experienced 1 AE; it was not related to the study drug
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) — 2 subjects on active treatment experienced 2 AEs and 1 subject on placebo experienced 1 AE; for 1 subject on active treatment and 1 subject on placebo it was possibly related to the study drug
Headache (Nervous system disorders) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 5 (7) — 4 subjects on active treatment experienced 6 AEs and one subject on placebo experienced 1 AE; none were related to the study drug
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) — 1 subject on active treatment experienced 1 AE and 2 subjects on placebo experienced 2 AEs; none were related to the study drug
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — 1 subject on active treatment experienced 1 AE; it was not related to the study drug
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — 2 subjects on active treatment experienced 2 AEs; they were not related to the study drug
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — 1 subject on active treatment experienced 1 AE; it was unlikely related to the study drug
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) — 2 subjects on placebo experienced 2 AEs
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — 1 subject on active treatment experienced 1 AE; it was not related to the study drug
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — 2 subjects on active treatment experienced 2 AEs; they were not related to the study drug
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — 1 subject on active treatment experienced 1 AE; it was not related to the study drug
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — 1 subject on placebo experienced 1 AE
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — 1 subject on active treatment experienced 1 AE; it was not related to the study drug
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) — 2 subjects on active treatment experienced 2 AEs and 1 subject on placebo experienced 1 AE; none were related to the study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI does not have the right to publish or otherwise present any results or data related to the study without an expressed written agreement from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT04632706/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04632706/SAP_001.pdf